CLINICAL TRIAL: NCT04953299
Title: Randomised Control Trial of Remote Access, Group-based Functional Imagery Training Versus NHS 12 Week Online Programme in the Community
Brief Title: Investigating Remote Access, Group-based Functional Imagery Training in the Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Plymouth (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Sarah Greene, Principal Investigator, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FITRCT
Record Dates: First submitted 2021-06-19; First posted 2021-07-07 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Weight Loss; Health Economics; Quality of Life
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Two groups of participants- one acts a control group and accesses the NHS 12 week programme the other group receives the FIT intervention.
Who Masked: Outcomes Assessor
Masking Description: The participants will not be masked to group allocation, data collection will be completed by a student apprentice blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Imagery training (Experimental): The FIT sessions will occur weekly for four weeks and last an hour per session. The sessions will be conducted over Zoom. Sessions will be facilitated by the PI who is trained in FIT, and attended by 4 participants.
  Interventions: Behavioral: Functional Imagery training
- Control (Active Comparator): The control condition will ask participants to complete the 12 week NHS weight loss plan.
  Interventions: Behavioral: NHS 12 week weight loss programme

INTERVENTIONS:
Behavioral: Functional Imagery training — Behavioural intervention focused upon motivation and reaching achievable goals.
  Arms: Functional Imagery training
Behavioral: NHS 12 week weight loss programme — The plan is designed to help individuals lose weight at a safe rate of 0.5kg to 1kg (1lb to 2lb) each week by sticking to a daily calorie allowance and introducing exercise.
  Arms: Control

SUMMARY:
The rise in obesity over the last two decades has led to an increased need to support individuals to lose weight but also reduce costs for healthcare settings. A review of group interventions for those with severe obesity concluded that group interventions are not only cost effective but also have good outcomes in terms of weight loss. A systematic review of individual and group based interventions for treating obesity found that group interventions were more effective but that the domain needed to be further explored.

Functional Imagery Training is a theoretically informed intervention that utilises client's intrinsic motivation to elicit effective behaviour change. It has drawn upon aspects of motivational interviewing and the use of imagery to develop an intervention that has been effective in many aspects including maintained weight loss when used on a 1:1 basis.

The investigators will conduct a Randomised Control Trial to test group-based delivery of FIT using the virtual platform Zoom versus the NHS 12 week online program as the current standard of what individuals seeking to lose weight can access independently.

DETAILED DESCRIPTION:
In England two thirds of the population are overweight, as defined by a body mass index (BMI) of 25 kg/m2 or more and nearly half of these have obesity as defined by a BMI of 30 kg/m-2 or more. Subsequently healthcare costs increase alongside the increasing prevalence of obesity and overweight with approximately 1.8% of the National Health Services (NHS) government budget and around 7.1% of all deaths being attributed to elevated BMI in 2014. Alongside the increased health risk associated with obesity, perceived quality of life declines also with increasing BMI. Tackling the obesity epidemic could therefore lead to better physical and mental health amongst a high proportion of the population.

The rise in obesity over the last two decades has led to an increased need to support individuals to lose weight but also reduce intervention costs. A review of group interventions for tier 3 services (severe obesity/ those with co-morbidities) found that group interventions are a cost effective method of treatment which demonstrate good results in terms of weight loss. Including the role of behaviour change in weight management is vital in ensuring the adoption and maintenance of new, long term skills which will help support maintaining weight loss.

Functional Imagery Training (FIT) is a theoretically informed intervention that utilises clients' intrinsic motivation and mental imagery to elicit effective behaviour change. It uses the well- established, person-centred approach of motivational interviewing. The mental imagery exercises are designed to strengthen motivation, consolidate plans for change, and build the person's confidence that they can succeed. Research demonstrates the emotive power of mental imagery and the shift from short-term rewards to longer term goals. Delivered face to face, one-to-one, FIT has been shown to elicit behaviour changes to support weight loss over a sustained period of 12 months. The investigators conducted a randomised controlled trial of one-to-one FIT compared to motivational interviewing which demonstrated those in the FIT group experienced greater weight loss at 6 months post-allocation compared to the motivational interview group and continued weight loss for the FIT group only at 12m, 6 months after intervention ended. There is a need to establish if FIT remains efficacious and cost-effective when delivered to groups.

The investigators will conduct a randomised control trial to test group-based delivery of FIT using the virtual platform Zoom. The current climate surrounding the increased need for remote-accessed services has allowed the investigators to explore the potential use of FIT online. There are many benefits to remote access interventions including reduced costs and travel time for the patients, more convenience and flexibility for patients and the reduced amount of clinic time for practitioners and patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* BMI over 30 kg/m2
* Access to an internet accessible device with camera and microphone facilities such as a smartphone, laptop, tablet or PC
* Access to weighing scales and a tape measure to self-report weight and waist measurements.

Exclusion Criteria:

* Current pregnancy
* Not fluent in English at a level that would allow them to participate in a group
* Not willing to be randomised
* Not willing to be part of a group
* Not able to complete baseline data
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) change | Change in BMI from baseline to 12 months
  kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared
waist circumference change | Change in waist circumference from baseline to 12 months
  Measured in centimetres

SECONDARY OUTCOMES:
EQ-5D-5L change (EuroQol-5D-5L) | Change in EQ-5D-5L score from baseline to 12 months
  Questionnaire score maximum 25, minimum 5, lower scores refer to better outcomes.
ICECAP-A change (ICEpop CAPability measure for Adults) | Change in ICECAP-A score from baseline to 12 months
  Questionnaire score, maximum 20 minimum 5, higher scores refer to better outcomes.
Health economics change | Change in service use from baseline to 12 months
  Descriptive score derived from a survey of service use

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Greene, Bsc, Ma, Principal Investigator — University of Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available including BMI, waist measurement, questionnaire responses and interview transcripts.
Time Frame: The data will be available once all the data has been analysed and submitted to a peer reviewed journal for publication. The full anonymised data set will then be available indefinitely.
Access Criteria: The anonymised data will be open-access.

REFERENCES:
- [Background] Solbrig L, Whalley B, Kavanagh DJ, May J, Parkin T, Jones R, Andrade J. Functional imagery training versus motivational interviewing for weight loss: a randomised controlled trial of brief individual interventions for overweight and obesity. Int J Obes (Lond). 2019 Apr;43(4):883-894. doi: 10.1038/s41366-018-0122-1. Epub 2018 Sep 5. PMID 30185920